CLINICAL TRIAL: NCT00246688
Title: Randomized, Multicenter, Prospective Two-arm, Open-label Phase II Study to Investigate the Efficacy and Safety of Two ZK219477 i.v. Infusions (3-hour Infusion of 16mg/m2 Versus 0.5-hour Infusion of 16 mg/m2) in Patients With Recurrent Ovarian Cancer Progressing During, or Within 6 Months of the End of Platinum-based Chemotherapy
Brief Title: Efficacy and Safety Study of ZK219477 in Patients With Recurrent Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 91447; 2005-000635-15 (EudraCT Number); 307970
Record Dates: First submitted 2005-10-28; First posted 2005-10-31 (Estimated); Last update posted 2015-12-31 (Estimated); Status verified 2015-12

CONDITIONS: Ovarian Neoplasms
MeSH Terms: conditions — Ovarian Neoplasms | interventions — sagopilone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sagopilone, 0.5 h infusion (Experimental): Subjects received one infusion (for 0.5 h) of sagopilone every 3 weeks at a dose of 16 mg/m2 (maximum up to 32 mg) for approximately 18 weeks
  Interventions: Drug: Sagopilone (BAY86-5302 , ZK219477)
- Sagopilone, 3 h infusion (Experimental): Subjects received one infusion (for 3 h) of sagopilone every 3 weeks at a dose of 16 mg/m2 (maximum up to 32 mg) for approximately 18 weeks
  Interventions: Drug: Sagopilone (BAY86-5302 , ZK219477)

INTERVENTIONS:
Drug: Sagopilone (BAY86-5302 , ZK219477) — 10.5 mg lyophilized sagopilone per vial

SUMMARY:
The purpose of this study is to determine if this epothilone leads to a response in patients with recurrent ovarian cancer that has progressed during, or in the last six months since a treatment of platinum-based chemotherapy. We also aim to look at the safety of the study drug and assess the impact of the infusion duration on tolerability.

DETAILED DESCRIPTION:
The study has previously been posted by Schering AG, Germany. Schering AG, Germany has been renamed to Bayer Schering Pharma AG, Germany.Bayer Schering Pharma AG, Germany is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:- Females aged 18 or over - Cancer of any of the following types: -- epithelial ovarian cancer -- peritoneal cavity cancer -- fallopian tube cancer - Up to 2 previous chemotherapies; the most recent must have been a platinum- containing therapy - Progression of disease or symptomatic relapse during, or within 6 months of previous therapy - 4 weeks or more since prior radiotherapy or chemotherapy - 3 weeks or more since prior immunotherapy - Adequate recovery from previous surgery, radiotherapy, and chemotherapy ( excluding alopecia) - Survival expectation of 3 months or more Exclusion Criteria: - More than 2 previous chemotherapies - Previous treatment with epothilones - Use of any investigational drug within 4 weeks of start of study treatment or inadequate recovery from any toxic effects of such therapy - Previous radiation to the whole pelvis - Symptomatic brain metastases requiring whole-brain irradiation - Active infection - Any other malignancy except: -- Non-melanoma skin cancer -- Carcinoma in situ of cervix -- Malignancy with treatment 5 or more years ago without relapse - Mixed mesodermal tumor - Prior hormone therapy for any malignancy in the previous month - Women of childbearing potential

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2005-11; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Proportion of responders | 18 weeks

SECONDARY OUTCOMES:
Duration of response | up to 1 year after LPLTV
Time to disease progression | up to 1 year after LPLTV
Number of participants with adverse events | Approximately 30 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer

REFERENCES:
- [Result] Rustin G, Reed N, Jayson GC, Ledermann JA, Adams M, Perren T, Poole C, Lind M, Persic M, Essapen S, Gore M, Calvert H, Stredder C, Wagner A, Giurescu M, Kaye S. A phase II trial evaluating two schedules of sagopilone (ZK-EPO), a novel epothilone, in patients with platinum-resistant ovarian cancer. Ann Oncol. 2011 Nov;22(11):2411-2416. doi: 10.1093/annonc/mdq780. Epub 2011 Mar 3. PMID 21372124
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/